CLINICAL TRIAL: NCT01728818
Title: Gemcitabine in Combination With the Oral Irreversible ErbB Inhibitor Afatinib Versus Gemcitabine Alone in Patients With Metastatic Pancreatic Cancer: an Explorative Randomized Phase II Trial
Brief Title: Afatinib as Cancer Therapy for Exocrine Pancreatic Tumours
Acronym: ACCEPT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PD Dr. med. Volker Heinemann (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, PD Dr. med. Volker Heinemann, Sponsor Delegated Person, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-004063-77
Record Dates: First submitted 2012-07-05; First posted 2012-11-20 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Focus of Study Instead
MeSH Terms: interventions — Gemcitabine; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Afatinib
- Arm B (Active Comparator)
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m² d1,8,15 q4weeks
  Arms: Arm A
Drug: Afatinib — 40mg flat dose, po, once daily
  Arms: Arm A
Drug: Gemcitabine — 1000 mg/m², d1,8,15 q4weeks
  Arms: Arm B

SUMMARY:
Single-agent gemcitabine is currently still regarded as one international standard of care for patients with advanced pancreatic cancer (Burris 1997 [4]). The oral EGFR tyrosine kinase inhibitor erlotinib received EMEA-approval for the treatment of patients with metastatic pancreatic cancer in January 2007.

In the pivotal phase III trial, the combination of gemcitabine plus erlotinib was associated with a statistically significant prolongation of OS (compared to single-agent gemcitabine), however, the absolute survival benefit was - for the overall study population - clinically moderate (median OS: 6.24 vs 5.91 months, 1-year OS rate: 23% vs 17%; HR = 0.82, p=0.038) (Moore 2007 [19]).

The recently presented FOLFIRINOX regimen shows enhanced activity in metastatic pancreatic cancer patients. This regimen is, however, limited to patients with good performance status (ECOG 0-1), no major comorbidity, age <75 years, and bilirubin <1.5 ULN (Conroy 2011 [6]). The majority of pancreatic cancer patients will therefore not be treated with this regimen.

Accordingly, novel treatment concepts are urgently needed in pancreatic cancer and pre-clinical data indicate an important role of the EGFR1/erbB2 receptor signalling in the pathogenesis of pancreatic adenocarcinoma (Yeh 2007 [24]). A recent publication (Larbouret 2010 [16]) indicates that the combination of cetuximab and trastuzumab induced superior antitumour activity in human pancreatic carcinoma xenografts compared to gemcitabine alone (see also Larbouret 2007 [15]). Furthermore, synergistic antitumour activity was observed when monoclonal antibodies directed against the EGFR1 and erbB2 were combined (Ben-Kasus 2009 [3]). Based on these data, there is a good rationale to further investigate the combined inhibition of the erbB family in pancreatic cancer patients.

Afatinib (BIBW 2992) is a novel irreversible EGFR1- and HER2 and HER4 inhibitor that is applied orally. The purpose of the present trial is to investigate the erbB family inhibition by afatinib in patients with metastatic pancreatic cancer.

In the planned trial, afatinib will be applied at the dose (40 mg/day) that was chosen for the randomised phase III trial (LUX 5 study) that investigates afatinib plus weekly paclitaxel (80mg/m2).

Presently there is also a phase I study ongoing that investigates the combination of afatinib with gemcitabine (ClinicalTrials.gov Identifier: NCT01251653 U10-2249-02 ). Possibly the data will be available once the study is ready to start. Otherwise a modification of the regimen will be planned once the respective data will be available.

In this trial, we integrate a translational project which may allow the identification of patients that primarily benefit from this novel treatment approach. The availability of tumour tissue- and blood samples from each patient is therefore an important inclusion criterion.

A 2:1 randomisation is chosen favouring the experimental arm since a large body of data is available on gemcitabine alone and since sufficient efficacy and toxicity data shall be gained in the experimental arm. In addition, the patients' motivation to take part in the trial will be greatly enhanced by a greater chance to receive the experimental agent.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in advance of any study-specific procedure
* Histologically (not cytologically) confirmed diagnosis of metastatic pancreatic adenocarcinoma (stage IV according to UICC 2009 classification: each T, each N, M1)
* Availability of tumour samples
* Informed consent that tumour- and blood samples are centrally collected and will serve for translational analyses according to the study protocol.
* Age >= 18 years
* ECOG 0-1
* Life expectancy at least 3 months
* No option for surgical resection or radiation in curative intent
* At least one measurable tumour lesion (CT-scan or MRI) according to RECIST Version 1.1
* Possibility of long-term follow-up
* Negative pregnancy test in fertile females
* Given legal capacity of the patient
* Adequate hepatic, renal and bone marrow function

Exclusion Criteria:

* Evidence of weight loss > 15% within one month
* Active brain metastases (stable for <28 days, symptomatic, or requiring concurrent steroids) or leptomeningeal disease. Patients who have received prior whole brain irradiation and whose brain metastases are stable according to the criteria above will not be excluded
* Previous gemcitabine treatment is allowed only if applied as monotherapy in the adjuvant setting and if the adjuvant single-agent gemcitabine chemotherapy was terminated at least 6 months before study entry
* Previous systemic treatment with chemotherapy or radiotherapy for locally advanced, non resectable or metastatic pancreatic cancer
* Radiotherapy within four weeks prior to randomization or radiation of target lesions
* Prior treatment with EGFR targeting therapies or treatment with EGFR- or HER2 inhibiting drugs within the past 4 weeks before start of therapy or concomitantly with this trial
* Hypersensitivity to afatinib or to gemcitabine or to any of the excipients or to compounds with similar chemical or biologic composition
* Contraindications against the use of gemcitabine
* Severe renal insufficiency (baseline creatinine clearance < 30 ml/mi)
* LDH elevated by > 2.5 ULN
* Severe hepatic dysfunction
* Any disease e. g. active infection, uncontrolled hypertension, clinically significant cardiovascular disease for example CVA (<= 6 months before study start), myocardial infarction (<= 6 months before study start), unstable angina, NYHA >= grade 2 CHF, arrhythmia requiring medication, metabolic dysfunction giving reasonable suspicion of a disease or condition that contra-indicates the use of the study drugs or puts the patient at high risk for treatment-related complications
* Significant or recent acute gastrointestinal disorders with diarrhoea as a major symptom e.g. Crohn's disease, malabsorption or CTC grade > 2 diarrhoea of any aetiology
* Pregnant or lactating females, non-effective contraception in men and women of childbearing potential (an effective contraceptive measure has a Pearl Index < 1)
* Any major surgery within the last 2 weeks before study entry
* Chemo- or immunotherapy within the past 4 weeks
* Treatment with an investigational drug in another clinical study within the past 28 days prior to the start of therapy or concomitantly with this study
* Any persisting toxicities which are deemed to be clinically significant from the previous therapy
* Patients with pre-existing interstitital lung disease
* Psychological, familial, social or geographic conditions that may prevent an adequate compliance with the study protocol
* Known or suspected alcohol- or drug abuse
* Patients unable to comply with the protocol
* Known hepatitis B infection, known hepatitis C infection or HIV carrier
* Requirement for treatment with any of the prohibited concomitant medications
* Any other malignancies within the last 5 years before study start, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-04; Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survial | approximately 36 months
  Overall Survival

SECONDARY OUTCOMES:
PFS | Approximately 36 months
  Progression-free survival (PFS)
Duration of response | approximately 36 months
  Duration of response
1 Year Survial | approximately 36 months
  One Year Survial
CA19-9 | approximately 36 months
  Biochemical tumour marker response (serum CA 19- 9)
Quality of life | approximately 36 months
  Evaluation of Quality of life with EORTC QLQ C-30 Questionaire
Toxicity | approximately 36 months
  Toxicity (NCI CTC-AE v4.0)
Staging | approximately 36 months
  All tumour assessments will be done by CT or MRI at 2-months intervals. One method of imaging will be kept consistent for each individual patient. All comparisons will be refrenced to baseline imaging (performed within 4 weeks prior to randomisation).

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, Professor, Principal Investigator — Medical Department III and Comprehensive Cancer Center
Locations (1):
- University of Munich, Munich, Germany

REFERENCES:
- [Derived] Weiss L, Heinemann V, Fischer LE, Gieseler F, Hoehler T, Mayerle J, Quietzsch D, Reinacher-Schick A, Schenk M, Seipelt G, Siveke JT, Stahl M, Vehling-Kaiser U, Waldschmidt DT, Dorman K, Zhang D, Westphalen CB, von Bergwelt-Baildon M, Boeck S, Haas M. Three-month life expectancy as inclusion criterion for clinical trials in advanced pancreatic cancer: is it really a valid tool for patient selection? Clin Transl Oncol. 2024 May;26(5):1268-1272. doi: 10.1007/s12094-023-03323-1. Epub 2023 Oct 4. PMID 37794220
- [Derived] Haas M, Waldschmidt DT, Stahl M, Reinacher-Schick A, Freiberg-Richter J, Fischer von Weikersthal L, Kaiser F, Kanzler S, Frickhofen N, Seufferlein T, Dechow T, Mahlberg R, Malfertheiner P, Illerhaus G, Kubicka S, Abdul-Ahad A, Snijder R, Kruger S, Westphalen CB, Held S, von Bergwelt-Baildon M, Boeck S, Heinemann V. Afatinib plus gemcitabine versus gemcitabine alone as first-line treatment of metastatic pancreatic cancer: The randomised, open-label phase II ACCEPT study of the Arbeitsgemeinschaft Internistische Onkologie with an integrated analysis of the 'burden of therapy' method. Eur J Cancer. 2021 Mar;146:95-106. doi: 10.1016/j.ejca.2020.12.029. Epub 2021 Feb 12. PMID 33588150
- See also: Homepage of the PancreasCenter at LMU Munich — http://www.klinikum.uni-muenchen.de/Pankreaszentrum-Muenchen/de/startseitenmeldungen/index.html